CLINICAL TRIAL: NCT05831202
Title: SEAL™IT: Saccular Endovascular Aneurysm Lattice System Interventional Pivotal Trial
Acronym: SEAL™IT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Galaxy Therapeutics INC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP0081
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Aneurysm
Keywords: Interventional Neurology; Intrasaccular Flow Diversion
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single arm (The SEAL™ Saccular Endovascular Aneurysm Lattice System) (Other): Prospective, US and OUS single-arm, multicenter, interventional study.
  Interventions: Device: The SEAL™ Saccular Endovascular Aneurysm Lattice System

INTERVENTIONS:
Device: The SEAL™ Saccular Endovascular Aneurysm Lattice System — All adult subjects between 22 and 80 years of age and presenting with an unruptured or ruptured saccular Wide Neck intracranial aneurysm with less or equal to 19 mm in its equatorial width (2mm-19mm range) that in the opinion of the Principal Investigator (PI) requires treatment and suitable candidate for intrasaccular flow diversion treatment, who meet all eligibility criteria, will be considered for study enrollment.

SUMMARY:
To establish the safety and effectiveness of the SEAL™ Saccular Endovascular Aneurysm Lattice system for the treatment of saccular intracranial aneurysms.

The data from this study will be used to support a premarket approval (PMA) submission.

DETAILED DESCRIPTION:
Prospective, United States (US) and Outside of the United States (OUS) single-arm, multicenter, interventional study. Patients presenting with evidence of Wide Neck unruptured or ruptured intracranial aneurysm (≤ 19 mm in widest diameter) requiring treatment will be enrolled into the study and treated using the SEAL™ System. Immediate post-procedure angiographic findings, clinical presentation, safety, and optional imaging follow-up for each subject will be collected at 24 hours or discharge, 3 months, 6 months, and required primary end point 12 months post-procedure. Digital subtraction angiography (DSA) at 12 months will be required imaging for the primary effectiveness endpoint assessment. After the PMA application, subjects follow up will continue annually for a total of five years post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. 22 to 80 years of age at the time of screening.
2. Unruptured aneurysm requiring endovascular treatment suitable for SEAL device and meet the American Heart Association (AHA) guidelines for management of unruptured aneurysm.5
3. Ruptured aneurysm A ruptured aneurysm is defined as a patient with computed tomography (CT), magnetic resonance imaging (MRI), or lumbar puncture (LP) evidence of Subarachnoid Hemorrhage (SAH) attributed to the index aneurysm within the last 60 days. Ruptured aneurysm may be included according to the following criteria:

   The subject is neurologically stable with no seizure at the onset of the SAH, not requiring External Ventricular Drain (EVD) placement prior to inclusion.
   * Hunt and Hess scale (HHS) of 2 or less at the time of treatment.
   * mRS of ≤2 prior to presentation or aneurysm rupture.
   * Meet the AHA guidelines for management of ruptured aneurysm.
4. The index intracranial aneurysm (IA) to be treated must include the following features:

   * Group A (primary analysis group): The Terminus/ bifurcation location:
   * 2 mm to 19 mm in equatorial aneurysm width wide neck aneurysm:
   * Absolute neck size ≥ 4mm and < 9mm AND Dome-to-Neck (DN) ratio ≥1 OR Dome- to-Neck (DN) ratio 1 to 2
   * Saccular morphology
   * Located in the anterior or posterior circulation
   * Group B (Expanded Indication): The Sidewall location:
   * 2 mm to 19 mm in equatorial aneurysm width wide neck aneurysm:
   * Absolute neck size ≥ 4mm and < 9mm AND Dome-to-Neck (DN) ratio ≥1 OR Dome- to-Neck (DN) ratio 1 to 2
   * Saccular morphology
   * Located in the anterior or posterior circulation
5. Aneurysm treatment does not require the preplanned use of any additional implanted devices.
6. Subject is able to maintain compliance with all aspects of screening, evaluation, treatment, and post-procedure follow-up schedule.
7. Baseline pre-procedure mRS of 0-2 for unruptured aneurysm and 0-2 prior to the SAH for the ruptured aneurysms.
8. Ability to obtain written informed consent document (ICD) subject or legally authorized representative in SAH subjects prior to the initiation of any study procedures.

Exclusion Criteria:

1. Aneurysm features unsuitable for endovascular treatment with an intrasaccular device such as fusiform, dissecting pseudo aneurysm, or mycotic aneurysm.
2. Aneurysms smaller than 2 mm and larger than 19 mm in dome width.
3. Patients with untreated multiple aneurysms [≥2mm]. Patient with multiple aneurysms, should have the none index aneurysms treated no less than 60 days prior to enrollment in the SEAL™ IT trial, ≤ 7mm, and not treated with flow diverter or stent assisted endovascular therapy.
4. Inability to access target aneurysm with microcatheter due to intracranial atherosclerosis, proximal or intracranial vessel tortuosity or poor aneurysm angle take-off.
5. Patients with two 360 degrees loops in the carotid or vertebral arteries.
6. Presence of vascular disease or other vascular abnormality that could prohibit access to index aneurysm such carotid stenosis or diminished caliber of the target artery.
7. Clinical, angiographic, or CT evidence of central nervous system (CNS) arterial vasculitis, Moyamoya disease, intracranial tumor (except small meningioma < 3 cm), or any other intracranial vascular malformations.
8. Patients with high risk for recurrent ischemic stroke due to previous history of ischemic stroke symptoms such as TIAs, minor, or major strokes within the past 60 days. Other stroke risk factors such as intracranial stenosis or atrial fibrillation.
9. Patients with hemodynamic or medical compromise due to medical comorbidities such as severe unstable congestive heart failure (ejection fraction <30%) or severe chronic obstructive pulmonary disease (COPD) requiring home oxygen.
10. Target index aneurysm that has been previously treated and contains devices, implants, or coils that could interfere with correct SEAL™ device placement.
11. Subject is pregnant or a lactating female (For females of child-bearing potential, a positive pregnancy test within 7 days of the day of procedure or refusal to use a medically accepted method of birth control for the duration of the study.
12. Currently on anticoagulation therapy or has a known blood dyscrasia, coagulopathy, or hemoglobinopathy.
13. Currently enrolled in another investigational study or post-market study that could affect the safety and efficacy of aneurysm treatment or interfere with the study follow-up schedule.
14. Presence of an acute life-threatening illness requiring treatment.
15. Life expectancy of < 5 years.
16. Subject has an uncontrolled co-morbid medical, neurological, or psychiatric condition, that would adversely affect participation in the study procedures and follow up.
17. Patient with chronic kidney disease (and not on dialysis) with creatinine > 2.0.
18. Subject with a known, uncontrolled hypersensitivity to iodine-based contrast dye, procedure related materials or medications, or device components^
19. Subject is a prisoner or member of other vulnerable population.
20. The subject that is in the opinion of the treating interventionalist is not suitable for the study.
21. Subjects with history of intracranial bleeding (SAH, SDH or ICH) within 90 days of the index aneurysm treatment.

    * Sensitivity to nickel is not specifically excluded, GTI performed ASTM F2129 testing recommended by the FDA in its 2015 and 2019 guiding documents. GTI results from the testing indicated that SEALTM meets the acceptance criteria that there is a high probability that the margin of safety against pitting (Eb-Er) is 200mV or higher, therefore, with high confidence, no further testing is required. The IFU contains the following precaution: "For patients with known hypersensitivity or allergic reaction to the implant components such as titanium or to nickel, use of the SEALTM System may lead to allergic reaction and user should counsel the patient on the device components".

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2030-09-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with successful aneurysm occlusion at 12 months | 12 Months
  Proportion of subjects with successful aneurysm occlusion at 12 months without parent artery stenosis or retreatment, as determined by independent core lab.

CONTACTS AND LOCATIONS:
Overall Officials: David Altschul, MD, Principal Investigator — Montefiore Health System; Brian Jankowitz, MD, Principal Investigator — JFK University Medical Center
Locations (6):
- United States (6):
  - Endeavor Health - Northwest Community Hospital, Arlington Heights, Illinois
  - Endeavor Health - Evanston Hospital, Evanston, Illinois
  - Endeavor Health- Edward Hospital, Naperville, Illinois
  - The Cooper Health System, Camden, New Jersey
  - NYU Langone Health, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York

IPD SHARING:
Plan to Share IPD: No